CLINICAL TRIAL: NCT02984826
Title: Muscle Strength in Shoulder and Neck Muscles in Adult Tension Type Headache Patients, and the Effect of Specific Strength Training
Brief Title: Muscle Strength in Shoulder and Neck Muscles in Tension Type Headache Patients. Effect of Specific Strength Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Bjarne Kjeldgaard Madsen, physiotherapist phd student, Danish Headache Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: H-3-2009-080
Record Dates: First submitted 2016-11-23; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-11

CONDITIONS: Tension-Type Headache
MeSH Terms: conditions — Tension-Type Headache | interventions — Resistance Training; Ergonomics; Posture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Strength training (Active Comparator): Intervention with specific strength training program runs for 10 weeks.
  Interventions: Other: Strength training
- Ergonomic and posture (Active Comparator): Intervention, the control group will be trained in ergonomics and posture.
  Interventions: Other: Ergonomic and posture

INTERVENTIONS:
Other: Strength training — The specific ST group trained and fulfilled a 10 week training diary. The ST consisted of 4 shoulder exercises. During the training the relative loading was progressively increased from 12 repetitions maximum (RM) (70% of maximal intensity) at the beginning to 8 RM (80 % of the maximal intensity). ST was performed with slow concentric and eccentric muscle contractions with resistance from the elastic bands.
  Arms: Strength training
Other: Ergonomic and posture — The control group was instructed in ergonomics and posture correction (EP). They were instructed to pay attention to their sitting posture, and how they used a computer or other working tools. Further they were asked to do a posture correction exercise 3 times a day with 10 repetitions. The EP were seen twice during the 10 week period, and had a phone call every 2 weeks. After 10 weeks they were instructed that they should stop the exercise but continue to be conscious of their ergonomics and sitting position.
  Arms: Ergonomic and posture

SUMMARY:
Background:

Tension Type Headache (TTH) is highly frequent and is of great socio-economic importance. Andersen et al. 2008 has shown that maximal muscle strength is reduced in women with trapezius myalgia. It is shown that specific strength training leads to prolonged pain relief.

Aim:Test: To investigate the impact of TTH on shoulder, and neck muscle strength in patients with TTH compared to healthy controls.

Intervention: To investigate the effect of specific strength training on patients with TTH compared with control group, receiving training in ergonomics.

Method: Test part. 60 tension headache patients, 30 healthy. Muscle testing of neck and shoulder. Testing conducted by blinded research assistant.

Intervention group: 60 patients with tension headache randomly assigned to the intervention group or control group. Intervention with specific strength training program runs for 10 weeks. The control group will be trained in ergonomics. 3 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* Tension-type headache(TTH), inclusion criteria were age between 18 and 65 years and for patients a diagnosis of TTH ≥8 headache days per month, and ≤3 migraine days per month according to ICHD-II -criteria.

Exclusion Criteria:

* Exclusion criteria were medication overuse headache (ICHD-II), previous whiplash or head trauma, other major physical or neurological diseases, depression, other mental illness, or being unable to understand and speak Danish. The patients were tested for cervicogenic headache according to Jull, et al 2007, and were excluded if the test was positive.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Headache frequency | Primary outcome headache frequency at (19-22 weeks)
  Frequency was calculated and analyzed as days with headache pr. month. primary outcome at follow up.(19-22 weeks)
Headache Duration | Primary outcome duration of pain at (19-22 weeks)
  The duration of the headache was registered in hours for each day with headache.

SECONDARY OUTCOMES:
Intensity of headache | Intensity of pain at (19-22 weeks)
  The intensity was registered on a 0-10 Numeric Rating Scale (NRS) where 0 is no pain, and 10 is worst possible pain. It was calculated as intensity mean/week and a mean for 4 weeks were produced
Medication intake | Medication intake at (19-22 weeks)
  Use of pain medicine was registered as days of medicine intake throughout the entire trial.

CONTACTS AND LOCATIONS:
Overall Officials: Bjarne K K Madsen, phd stud., Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center Rigshospitalet - Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Madsen BK, Sogaard K, Andersen LL, Tornoe B, Jensen RH. Efficacy of strength training on tension-type headache: A randomised controlled study. Cephalalgia. 2018 May;38(6):1071-1080. doi: 10.1177/0333102417722521. Epub 2017 Jul 27. PMID 28750588